CLINICAL TRIAL: NCT01132131
Title: Use of Standardized Delegation Form in Diagnosing and Treating Acute Cystitis in Primary Care Facilities.
Brief Title: Management of Urinary Tract Infections in Primary Care Facilities.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Oslo (Other)
Responsible Party: Principal Investigator, Marianne Bollestad, Md, University of Oslo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010/486
Record Dates: First submitted 2010-05-20; First posted 2010-05-27 (Estimated); Last update posted 2012-02-02 (Estimated); Status verified 2012-02

CONDITIONS: Urinary Tract Infection
Keywords: Urinary tract infection; Cystitis; Bacteruria
MeSH Terms: conditions — Urinary Tract Infections; Cystitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Delegation form (Active Comparator)
  Interventions: Other: Delegation form
- Regular doctor's consultation (Active Comparator)
  Interventions: Other: Delegation form

INTERVENTIONS:
Other: Delegation form — The study aims to compare the use of a delegation form to identify patient's who qualify for antibiotic treatment for suspected acute cystitis with a regular doctor's consultation. The key outcomes are lack of bacteruria and symptoms of UTI at followup times.

SUMMARY:
The Emergency Ward Center in Oslo has the last two years used a questionnaire to identify patients who qualify for treatment of acute cystitis by the use of a delegation form.

The aim of the study is to evaluate this practice, the primary objective being to evaluate if in a selected patient group the treatment outcome after identifying patients with probable acute cystitis by delegation form will be as good or better than the treatment received after a regular doctor's consultation.

The planned study will also investigate which symptoms, signs and laboratory findings that coincide with significant bacteruria.

The reference standard will be a microbiological culture of every patients urine.

ELIGIBILITY:
Inclusion Criteria:

* Females 16-55 years
* Dysuria
* Increased frequency of urination

Exclusion Criteria:

* Pregnant
* Breastfeeding child < 1 month of age
* Diabetes
* Kidney disease
* Fever
* Poor general condition
* Backpain
* Abdominal pain
* Increased amount of vaginal secretions
* Vaginal itching or pain
* Urinary tract infection in the last four weeks
* Use of urinary catheter in the last four weeks
* Symptoms lasting more than seven days
* Ongoing antibiotic treatment
* Allergy to penicillin
* Use of the medicine Probecid

Ages: 16 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 443 (Actual)
Dates: Start 2010-08; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Number of patients who are clinically and bacteriologically free of symptoms of urinary tract infection. | 6 days after start of treatment.
  The antibiotic treatment given will be of three days length.
Number of patients who are clinically and symptomatologically free of symptoms. | 10 days after start of treatment
  The antibiotic treatment will be of three days length

CONTACTS AND LOCATIONS:
Overall Officials: Morten Lindbaek, Md PhD, Study Director — University of Oslo
Locations (1):
- Legevakten i Oslo, Oslo, Oslo County, Norway

REFERENCES:
- [Derived] Bollestad M, Grude N, Lindbaek M. A randomized controlled trial of a diagnostic algorithm for symptoms of uncomplicated cystitis at an out-of-hours service. Scand J Prim Health Care. 2015 Jun;33(2):57-64. doi: 10.3109/02813432.2015.1041827. Epub 2015 May 11. PMID 25961367